CLINICAL TRIAL: NCT02977286
Title: Impact of Naloxegol on Prevention of Lower GI Tract Paralysis in Critically Ill Adults Initiated on Scheduled Intravenous Opioid Therapy: A Randomized, Double-Blind, Placebo-Controlled, Phase II, Single-Center, Proof of Concept Study
Brief Title: Naloxegol to Prevent Lower Gastrointestinal Paralysis in Critically Ill Adults Administered Opioids
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11200
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — naloxegol; Dioctyl Sulfosuccinic Acid; Sennosides; Tablets; Polyethylene Glycols; polyethylene glycol 3350; Bisacodyl; Suppositories; magnesium citrate; methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naloxegol Oral Tablet (Experimental): Intervention: Naloxegol 25 mg (or 12.5 mg) tablet po (enteral) daily AND Docusate Sodium 100mg Oral Capsule twice daily AND Study laxative protocol daily [that may include Senna 217 mg Oral Tablet, Polyethylene Glycols (Miralax), Magnesium Citrate Oral Liquid Product (Citromag), Bisacodyl 10 mg Suppository (Dulcolax) and Methylnaltrexone (Relistor)] until one of the following:
  1. Adverse event potentially attributable to the study drug.
  2. Use of Relistor.
  3. Scheduled opioid therapy is stopped for ≥ 24 hours and participant has ≥ 1 SBM since enrollment.
  4. The participant has been administered 10 days of study medication.
  5. The participant is discharged from the ICU.
  6. The participant requires the initiation of a strong CYP3A4 inhibitor medication.
  Other Name: Movantik
  Interventions: Drug: Naloxegol Oral Tablet; Drug: Docusate Sodium 100 Mg oral capsule [Colace]; Drug: Senna 217 Mg Oral Tablet; Drug: Polyethylene Glycols; Drug: Bisacodyl 10 mg Suppository; Drug: Magnesium Citrate Oral Liquid Product; Drug: Methylnaltrexone
- Placebo Oral Tablet (Placebo Comparator): Intervention: Placebo tablet po (enteral) daily AND Docusate Sodium 100 mg Oral Capsule twice daily AND Study laxative protocol daily [that may include Senna 217 mg Oral Tablet, Polyethylene Glycols (Miralax), Magnesium Citrate Oral Liquid Product (Citromag), Bisacodyl 10 mg Suppository (Dulcolax) and Methylnaltrexone (Relistor)] until one of the following:
  1. Adverse event potentially attributable to the study drug.
  2. Use of Relistor.
  3. Scheduled opioid therapy is stopped for ≥ 24 hours and participant has ≥ 1 SBM since enrollment.
  4. The participant has been administered 10 days of study medication.
  5. The participant is discharged from the ICU.
  6. The participant requires the initiation of a strong CYP3A4 inhibitor medication.
  Other Name: AstraZeneca provided Movantik placebo
  Interventions: Drug: Placebo Oral Tablet; Drug: Docusate Sodium 100 Mg oral capsule [Colace]; Drug: Senna 217 Mg Oral Tablet; Drug: Polyethylene Glycols; Drug: Bisacodyl 10 mg Suppository; Drug: Magnesium Citrate Oral Liquid Product; Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Naloxegol Oral Tablet — Naloxegol Oral Tablet 25 mg (or 12.5 mg) po (enteral) daily
  Other Names: Movantik
  Arms: Naloxegol Oral Tablet
Drug: Placebo Oral Tablet — Placebo Oral Tablet po (enteral) twice daily
  Other Names: Official AstraZeneca placebo for Movantik
  Arms: Placebo Oral Tablet
Drug: Docusate Sodium 100 Mg oral capsule [Colace] — Docusate Sodium 100 mg po (enteral) twice daily
  Other Names: Colace
Drug: Senna 217 Mg Oral Tablet — Senna 127 mg oral tablet daily if no spontaneous bowel movement >/=3 days after scheduled opioid initiation; increase to two senna 127 mg tables if no no spontaneous bowel movement >/=4 days after scheduled opioid initiation. Repeat two senna 127 mg tablets if no spontaneous bowel movement >/=5 days after scheduled opioid initiation. Repeat two senna 127 mg tablets if no spontaneous bowel movement >/=6 days after scheduled opioid initiation.
  Other Names: Senokot
Drug: Polyethylene Glycols — Polyethylene Glycols 17 g daily if no spontaneous bowel movement >/=3 days after scheduled opioid initiation; increase to 34 g daily if no spontaneous bowel movement >/=4 days after scheduled opioid initiation. Repeat 34 g daily if no spontaneous bowel movement >/= 5 days after scheduled opioid initiation. Repeat 34 g daily if no spontaneous bowel movement >/= 6 days after scheduled opioid initiation.
  Other Names: Miralax
Drug: Bisacodyl 10 mg Suppository — Insert one suppository if no spontaneous bowel movement >/=4 days after scheduled opioid initiation. Repeat if no spontaneous bowel movement >/= 5 days after scheduled opioid initiation. Repeat if no spontaneous bowel movement >/= 6 days after scheduled opioid initiation.
  Other Names: Dulcolax
Drug: Magnesium Citrate Oral Liquid Product — Administer one 10 oz bottle if no spontaneous bowel movement >/= 5 days after scheduled opioid initiation.
  Other Names: Citromag
Drug: Methylnaltrexone — Administer 8 mg or 16 mg (depending on subject's weight) subcutaneously x 1 if no spontaneous bowel movement >/= 6 days after scheduled opioid initiation, consult surgery/gastroenterology and discontinue study medication.
  Other Names: Relistor

SUMMARY:
This study evaluates the addition of naloxegol (Movantik) to a laxative protocol in critically ill adults requiring scheduled opioid (e.g. fentanyl) therapy. Half of the participants will receive naloxegol and a laxative protocol and half the participants will receive a placebo and a laxative protocol.

DETAILED DESCRIPTION:
Among the more than 5 million adults who are admitted to the ICU each year in the USA, most have pain and thus receive a pain (analgesic) medication called an opioid. Opioid use in critically ill adults continues to increase given the greater awareness of untreated pain in the ICU and that an opioid-first approach be used to optimize patient safety and comfort and improve tolerance with breathing machines (i.e. mechanical ventilation). Similar to constipation, paralysis of the lower gastrointestinal (GI) tract is defined as the inability to pass stool due to impaired gut movement, and is a common effect of opioid use in the critically ill. Lower GI tract paralysis may lead to nausea, vomiting, aspiration, compromise the ability to administer tube feeds (enteral nutrition), an increase abdominal pain, delirium and delay getting off mechanical ventilation. One recent randomized study found that aggressive use of laxatives to prevent lower GI tract paralysis in critically ill adults was associated with lower daily organ dysfunction [as measured by the Sequential Organ Failure Assessment (SOFA) score]. The lower GI tract paralysis that occurs in the critically ill often responds poorly to laxative medication therapy (e.g., senna, bisacodyl, lactulose). While stool softener medications like docusate are routinely administered to patients on opioids, laxative-based protocols are frequently not initiated in the ICU until signs of lower GI tract paralysis start to appear. There is therefore an important and unmet need for a safe and efficacious medication to prevent lower GI tract paralysis in critically ill adults who are initiated on opioid therapy. Naloxegol (Movantik) is a naloxone-like drug that blocks the effect of opioids on the opioid µ receptor in the gut but is not absorbed in the brain (and therefore does not block the pain effects of opioids). Naloxegol is currently approved by the Food and Drug Administration (FDA) for the treatment of opioid-induced constipation (OIC) in non-ICU patients receiving scheduled moderate to high dose opioids for the treatment of chronic non-cancer pain. Naloxegol has a mechanism of action, efficacy, convenience of administration, and safety profile that make it an ideal candidate for use as a preventative medication for lower GI tract paralysis in critically ill adults receiving scheduled opioid therapy. The investigators propose a pilot study in which they will test the hypothesis that naloxegol (versus placebo) will reduce the time to the first spontaneous bowel movement (SBM) that an ICU patient has, that it will prevent lower GI tract paralysis in critically ill adults initiated on scheduled IV opioid therapy, and its use will not result in side effects that are concerning to doctors or patients. The investigators will randomize 36 critically ill ICU patients (18 in each arm) to receive naloxegol [25mg or 12.5mg (in patients with a creatinine clearance ≤ 60ml/min)] or placebo. This pilot study will provide valuable information to help guide future, larger studies evaluating the role of naloxegol in critically ill adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to an ICU
* Expected to require admission to an ICU for ≥ 48 hours
* Intravenous opioid administration in the prior 24 hours of ≥ 100 mcg fentanyl equivalents

Exclusion Criteria:

* Scheduled use of an opioid ≥ 10 mg morphine equivalents per day in the week prior to ICU admission
* History of constipation (≤ 2 SBM per week and current use of stool softener or laxative therapy) prior to ICU admission
* Current scheduled use of a medication affecting gastric motility
* Current use of a medication known to be a strong CYP3A4 inhibitor
* History of a neurologic condition that may affect the permeability of the blood-brain barrier
* Acute GI condition (e.g., clinical evidence of acute fecal impaction/complete obstruction, acute surgical abdomen, acute GI bleeding)
* Condition affecting GI motility or function (e.g. inflammatory bowel disease requiring immunosuppressive therapy, symptomatic Clostridium difficile, active diverticular disease, surgery on the colon or abdomen within 60 days of ICU admission)
* Current use of total parenteral nutrition
* Administration of enteral nutrition through a jejunal tube
* Severe hepatic dysfunction
* Endstage renal disease defined as either i. calculated creatinine clearance ≤ 10ml/min or ii. Any current use of renal replacement therapy
* Inability to enroll in study and initiate study medication within 48 hours of the patient begin first initiated on scheduled IV opioid therapy after ICU admission
* Unreliable method for enteral, gastric and/or oral medication administration (e.g., no feeding tube, nasogastric tube is on suction)
* Current or previous use of an opioid antagonist agent (e.g., naloxegol, methylnaltrexone) in the past 30 days
* Pregnant or actively lactating females
* Current participation in another interventional clinical study
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Garpestad, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869
- [Background] de Azevedo RP, Freitas FG, Ferreira EM, Pontes de Azevedo LC, Machado FR. Daily laxative therapy reduces organ dysfunction in mechanically ventilated patients: a phase II randomized controlled trial. Crit Care. 2015 Sep 16;19(1):329. doi: 10.1186/s13054-015-1047-x. PMID 26373705

RESULTS

PARTICIPANT FLOW:
Groups:
- Naloxegol Oral Tablet: Intervention: Naloxegol 25 mg (or 12.5 mg) tablet po (enteral) daily AND Docusate Sodium Oral Capsule twice daily AND Study laxative protocol daily [that may include Senna Oral Tablet, Polyethylene Glycols, Magnesium Citrate Oral Liquid Product, Bisacodyl Suppository and Methylnaltrexone] until one of the following:
  1. Adverse event potentially attributable to the study drug.
  2. Use of Relistor.
  3. Scheduled opioid therapy is stopped for ≥ 24 hours and participant has ≥ 1 SBM since enrollment.
  4. The participant has been administered 10 days of study medication.
  5. The participant is discharged from the ICU.
  6. The participant requires the initiation of a strong CYP3A4 inhibitor medication.
  Other Name: Movantik
Period: Overall Study
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (23) | 64 (11) | 57 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
BMI [Mean (Standard Deviation); unit: kg/m2] | 40 (13) | 35 (16) | 38 (14)
APACHE-II: Acute Physiology and Chronic Health Evaluation (version II) [Mean (Standard Deviation); unit: units on a scale] — APACHE II score is a general measure of disease severity based on current physiologic measurements, age and previous health conditions. Minimal score is 0, maximum is 71.
  Higher value suggests worse outcome.
  units on a scale | 20 (6) | 19 (7) | 19.5 (6.5)
SOFA score: Sequential Organ Failure Assessment Score [Mean (Standard Deviation); unit: units on a scale] — SOFA score is used to track a patient's status, usually during a admission to an Intensive Care Unit. This score tracks patient's organ function or rate of failure. Score is 0 to 24. Higher score is worse, with more organ failure.
  units on a scale | 8 (4) | 6 (2) | 7 (3)
Hours in ICU before enrollment [Mean (Standard Deviation); unit: hours] | 50 (21) | 44 (21) | 48 (22)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Spontaneous Bowel Movement (SBM) Administration
Description: Time to first spontaneous bowel movement during ICU admission after randomization
Time Frame: First occurrence after study randomization during period of ICU admission or a maximum of 10 ICU days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
hours | 41 (25) | 33 (25)

2. Secondary Outcome: Time to First Spontaneous Bowel Movement (SBM)
Description: Time to first spontaneous bowel movement during the ICU admission after opioid initiation
Time Frame: First occurrence after initiation of IV opioid therapy during period of ICU admission or a maximum of 10 ICU days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
hours | 52 (28) | 49 (38)

3. Secondary Outcome: ICU Days Without a SBM
Description: Measured ICU days that subjects did not have a SBM
Time Frame: During period of ICU admission or a maximum of 10 ICU days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Naloxegol Oral Tablet: Intervention: Naloxegol 25 mg (or 12.5 mg) tablet po (enteral) daily AND Docusate Sodium 100mg Oral Capsule twice daily AND Study laxative protocol daily [that may include Senna 217 mg Oral Tablet, Polyethylene Glycols (Miralax), Magnesium Citrate Oral Liquid Product (Citromag), Bisacodyl 10 mg Suppository (Dulcolax) and Methylnaltrexone (Relistor)] until one of the following:
  1. Adverse event potentially attributable to the study drug.
  2. Use of Relistor.
  3. Scheduled opioid therapy is stopped for ≥ 24 hours and participant has ≥ 1 SBM since enrollment.
  4. The participant has been administered 10 days of study medication.
  5. The participant is discharged from the ICU.
  6. The participant requires the initiation of a strong CYP3A4 inhibitor medication.
  Other Name: Movantik
  .
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
Days | 2 (3) | 2 (2)

4. Secondary Outcome: Occurrence of Lower GI Tract Paralysis (≥3 Days Without a SBM)
Description: Measurement is the number of subjects in each group having this occurrence of lower GI tract paralysis during time frame
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Count of Participants; unit: Participants
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
Participants | 2 | 3

5. Secondary Outcome: Average Daily Opioid Requirement [in IV Fentanyl Equivalents (mcg Per Day)]
Description: Average daily opioid requirement is converted to IV fentanyl equivalent listed in mcg per day
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Mean (Inter-Quartile Range); unit: mcg per day
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
mcg per day | 1420 [65 to 3548] | 1600 [1105 to 2382]

6. Secondary Outcome: Number of Patients With Loose and Unformed or Liquid SBM
Description: Consistency of SBM is characterized in one of 4 categories: hard and formed, soft but formed, loose and unformed, and liquid. The number listed in the results section is the number of patients who had either loose or liquid SBM (as opposed to hard or soft formed).
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Count of Participants; unit: Participants
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
Participants | 5 | 6

7. Secondary Outcome: Number of Patients That Required Use of the Study Laxative Protocol
Description: A 4-step laxative protocol was initiated when there was no spontaneous bowel movement greater than or equal to 3 days time. Data collected on study laxative protocol included any use as well as the highest level needed.
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Number; unit: participants
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
participants | 5 | 4

8. Secondary Outcome: Percentage of Daily Goal Reached for Enteral Nutrition Administration
Description: Enteral nutrition is assessed as daily volume in mL and the reported measure is the percentage of daily goal of enteral nutrition met.
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Mean (Standard Deviation); unit: percentage of daily goals met
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
percentage of daily goals met | 54 (34) | 51 (29)

9. Secondary Outcome: Daily Fluid Balance
Description: Daily fluid balance measured in mL is the 24 hours ins and outs
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Mean (Inter-Quartile Range); unit: mL
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
mL | -338 [-747 to -102] | -210 [-660 to -208]

10. Secondary Outcome: Daily Maximal Pain Scale Score
Description: Based on the highest daily Visual Analogue Scale-10 or Clinical Pain Observation tool assessment.
  VAS-10 is Visual Analogue Scale which uses a nurse-administered 10 point rating scale. A measurement of 0-1 is minimal pain. A measurement of 10 is severe pain.
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Placebo Oral Tablet: Intervention: Placebo tablet po (enteral) daily AND Docusate Sodium 100 mg Oral Capsule twice daily AND Study laxative protocol daily [that may include Senna 217 mg Oral Tablet, Polyethylene Glycols (Miralax), Magnesium Citrate Oral Liquid Product (Citromag), Bisacodyl 10 mg Suppository (Dulcolax) and Methylnaltrexone (Relistor)] until one of the following:
  1. Adverse event potentially attributable to the study drug.
  2. Use of Relistor.
  3. Scheduled opioid therapy is stopped for ≥ 24 hours and participant has ≥ 1 SBM since enrollment.
  4. The participant has been administered 10 days of study medication.
  5. The participant is discharged from the ICU.
  6. The participant requires the initiation of a strong CYP3A4 inhibitor medication.
  Other Name: AstraZeneca provided Movantik placebo
  ation.
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
score on a scale | 0 [0 to 3] | 0 [0 to 0]

11. Secondary Outcome: Daily Maximal Sedation Assessment Scale (SAS) Score
Description: The Sedation Assessment Scale is rated 1 to 7. Score of 7 is dangerous agitation. Score of 1 is unarousable. Score of 2 is very sedated. The presence of coma is based on the every 4 hour sedation agitation score scale (SAS) assessment. A score of 1 or 2 any time during the day represents that a coma is present. A score of 3-7 represents a subject with no coma present.
  Results listed here is days without coma (SAS score of 3-7)
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
days | 3 [1 to 3] | 7 [4 to 7]

12. Secondary Outcome: Daily Presence of Delirium Using the Intensive Care Delirium Screening Checklist (ICDSC)
Description: Measures as days without delirium with daily presence of delirium assessed using the Intensive Care Delirium Screening Checklist (ICDSC)
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Median (Inter-Quartile Range); unit: days without delirium
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
days without delirium | 5 [4 to 6] | 6 [4 to 7]

13. Secondary Outcome: Occurrence of Lower GI Tract Paralysis Requiring GI/Surgical Consultation
Description: Number of patients with GI tract paralysis requiring Gastroenterology service or Surgical service consultation
Time Frame: From randomization to ICU discharge or a maximum of 10 ICU days
Measure: Count of Participants; unit: Participants
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

14. Secondary Outcome: Days Without Mechanical Ventilation Support for Duration of ICU Stay
Description: Measure is days without mechanical ventilation for duration of ICU stay as expressed as median and inter-Quartile Range
Time Frame: From ICU admission to ICU discharge or a maximum of 10 ICU days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
days | 0.5 [0.2 to 5] | 1 [0.3 to 3]

15. Secondary Outcome: Abdominal Pressure Measurement
Description: On days when the patient had a urinary catheter in place for clinical reasons, a bladder pressure transducer was inserted and abdominal pressure was measured. The average daily maximum pressure score for each group is reported.
Time Frame: From randomization to ICU discharge (or removal of foley catheter) or a maximum of 10 ICU days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 4
mmHg | 10 (4) | 13 (5)

16. Secondary Outcome: Time to First Episode of Diarrhea
Description: The number of patients in each group with > or equal to 1 episode of diarrhea after initiation of study drug. The time to first episode of diarrhea was measured in hours.
Time Frame: Study drug initiation to first episode of diarrhea in hours.
Population: Number of patients in each group with > or equal to 1 episode of diarrhea.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 4 | 4
hours | 40 [19 to 66] | 109 [48 to 169]

17. Secondary Outcome: Daily Difference in the Pre-dose and Post-dose Clinical Opioid Withdrawal Scale (COWS) Score
Description: Patients were evaluated 1 hour before and 2 hours after the administration of each dose of study medication using the Clinical Opioid Withdrawal Scale (COWS). COWS is used to help determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. The COWS score ranges from 0-36+. A score of 0 is no active opioid withdrawal. A score of 5-12 is mild; 13-24 is moderate; 25-36 is moderately severe and more than 36 is severe opioid withdrawal.
Time Frame: One hour before the daily study drug administration and 2 hours after the daily study drug administration
Measure: Mean (Standard Deviation); unit: Difference of COWS score
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 6 | 6
Difference of COWS score | -0.1 (1.3) | 0.2 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject during the period from time of study enrollment (i.e. randomization) to ICU discharge, death or 10 days of study drug administration (whatever comes first).
Arm/Group | Naloxegol Oral Tablet | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxegol Oral Tablet (N=6) | Placebo Oral Tablet (N=6)
Diarrhea (Gastrointestinal disorders) | 4 | 4 — Diarrhea defined where greater than or equal to 3 loose or watery stools (Bristol stool scale score of 6 or 7) in a 24 hour period.

LIMITATIONS AND CAVEATS:
Limitations: One-third of the planned participants were enrolled, thus the study is substantially underpowered. Our results do not apply to non-medical patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT02977286/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT02977286/SAP_001.pdf
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT02977286/ICF_002.pdf